CLINICAL TRIAL: NCT03365323
Title: Diagnosis of Periprosthetic Joint Infection and the Common Pathogens, Durg-resistance in Periprosthetic Joint Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Jianhao, The clinical professor of arthritis clinic and research center, Peking University People's Hospital
Other Study IDs: PKUPHACRC3
Record Dates: First submitted 2017-11-25; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Arthropathy of Hip; Arthropathy of Knee
Keywords: Periprosthetic Joint Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Collected lab examinations included blood routine test, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), synovial leukocyte counts, as well as microorganisms isolated from periprosthetic tissues and articular fluid.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- infectious group: Patients who met the criteria according of Periprosthetic Joint Infection were identified as the infectious group.
  Interventions: Other: Periprosthetic Joint Infection
- non-infectious group: Patients who didn't meet the criteria according of Periprosthetic Joint Infection were identified as the non-periprosthetic joint infection group.
  Interventions: Other: Non-Periprosthetic Joint Infection

INTERVENTIONS:
Other: Periprosthetic Joint Infection — Periprosthetic Joint Infection is diagnosed according to the diagnosing criteria from the Workgroup of the Musculoskeletal Infection Society.
  Groups: infectious group
Other: Non-Periprosthetic Joint Infection — PJI can not be diagnosed for the lack of clinical evidence according to the diagnosing criteria from the Workgroup of the Musculoskeletal Infection Society.
  Groups: non-infectious group

SUMMARY:
This retrospective study aims to improve the diagnosis of PJI as well as to identify microorganisms causing periprosthetic joint infection (PJI) and the drug-resistant spectrum

DETAILED DESCRIPTION:
160 patients who underwent revision or re-revision total hip or knee arthroplasty for different reasons in our institution were recruited from August 2013 to August 2016. 80 patients meet the criteria of PJI from the muscle and skeletal muscle Association (MSIS) are divided to the infection group, another 80 patients are divided into the non-infection group.

Medical and demographic data were recorded. Collected lab examinations included blood routine test, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), synovial leukocyte counts, Receiver Operating Characteristic Curve-Area Under Curve (ROC-AUC) analysis will be used to evaluate the specific and sensitivity of diagnosis index. Moreover,microorganisms isolated from periprosthetic tissues and articular fluid. Postoperatively, the prosthesis was sent for ultrasound sonication. The sonicate extraction, implant surrounding tissue and synovium were sent for microbiologic culture, and the implant-surrounding-tissue were also sent for pathological examination. The isolated strains and drug-resistance rate for each bacterium for different antibiotics were presented.

ELIGIBILITY:
Inclusion Criteria:

* patient who underwent revision or re-revision total hip or knee arthroplasty for different reasons in our institution

Exclusion Criteria:

1. Patients who refused to join the trial group;
2. Revision total hip/knee replacement for periprosthetic fracture;
3. patients who missed some of important examination;
4. Revision total hip/knee replacement for metal sensitivity;
5. Revision total hip/knee replacement for the last period of second-stage revision;
6. Patient who underwent revision with RA or other inflammatory disease.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent revision or re-revision total hip or knee arthroplasty for different reasons in our institution
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation the specific and sensitivity of CRP | within 4 weeks before the operation
  To test the specifity and sensitivity of CRP
Evaluation the specific and sensitivity of ESR | within 4 weeks before the operation
  To test the specifity and sensitivity of ESR
Evaluation the specific and sensitivity of synovial leukocyte counts | within 4 weeks before the operation
  To test the specifity and sensitivity of synovial leukocyte counts

SECONDARY OUTCOMES:
Microorganisms identification and the | within 4 weeks before the operation
  Identify microorganisms causing periprosthetic joint infection (PJI) as well as the drug-resistant spectrum.
Drug-resistant spectrum. | within 4 weeks before the operation
  Identify the drug-resistant spectrum of the microorganisms.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, Principal Investigator — arthritis and clinic and research center

IPD SHARING:
Plan to Share IPD: No